CLINICAL TRIAL: NCT01738646
Title: Phase II Study of Bevacizumab and Vorinostat for Recurrent WHO Grade IV Malignant Glioma Patients
Brief Title: Ph II SAHA and Bevacizumab for Recurrent Malignant Glioma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024983
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-11

CONDITIONS: Recurrent Glioblastoma Multiforme; Malignant Glioma; Adult Brain Tumor
Keywords: vorinostat; SAHA; bevacizumab; AVASTIN; malignant glioma; GBM; glioblastoma multiforme; brain tumor
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Vorinostat; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat & Bevacizumab (Experimental): Patients will be administered bevacizumab every 2 weeks and vorinostat will be taken on days 1-7 and 15-21 of each 28-day cycle at 400 mg per day.
  Interventions: Drug: Vorinostat; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vorinostat
  Other Names: SAHA
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
It has been shown that bevacizumab has significant anti-tumor activity in patients with recurrent glioblastoma multiforme. Vorinostat has modest anti-tumor activity against malignant glioma and can enhance the action of both chemotherapy and anti-angiogenics. Patients will be treated with a combination of bevacizumab and vorinostat.

DETAILED DESCRIPTION:
There is no effective therapy for patients with recurrent glioblastoma multiforme (GBM) hence such patients remain a major unmet need in oncology. The investigators have recently demonstrated that bevacizumab (BV), a humanized monoclonal antibody against vascular endothelial growth factor, has significant anti-tumor activity among recurrent glioblastoma multiforme patients. Vorinostat has modest anti-tumor activity against malignant glioma and can potentiate the action of both chemotherapy and anti-angiogenics. The current study is designed to evaluate the anti-tumor activity of vorinostat when combined with BV among recurrent glioblastoma multiforme patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* An interval of at least 4 weeks between prior surgical resection or one week from stereotactic biopsy.
* An interval of at least 12 weeks from the end of prior radiotherapy unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there is biopsy-proven tumor progression
* An interval of at least 4 weeks from prior chemotherapy [6 weeks for nitrosoureas, 1 week for daily administered chemotherapy (metronomic dosing)] or investigational agent unless the patient has recovered from all anticipated toxicities associated with that therapy.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* Hematocrit ≥ 29%, hemoglobin ≥ 9, absolute neutrophil ≥1,500 cells/microliter, platelets ≥ 100,000 cells/microliters.
* Serum creatinine, serum glutamic oxaloacetic transaminase(SGOT) and bilirubin < 1.5 times upper limit of normal.
* Signed informed consent approved by the Institutional Review Board prior to patient entry.
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are stable grade 1.
* If sexually active, patients will take contraceptive measures for the duration of the treatments. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation, hysterectomy, vasectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD).

Exclusion Criteria:

Disease-specific exclusions

* More than 2 prior episodes of disease progression
* Prior therapy with histone deacetylase inhibitors; valproic acid is not permitted and patients previously treated with valproic acid must be off valproic acid for at least 30 days prior to initiation of study medication
* Prior bevacizumab therapy
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Active infection requiring intravenous antibiotics
* Severe hepatic insufficiency, active viral hepatitis or HIV infection
* Requires therapeutic anti-coagulation with warfarin

General medical exclusions

Subjects meeting the following criteria are ineligible for study entry:

* Inability to comply with study and/or follow-up procedures

Bevacizumab-specific exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either:

  * Urine protein:creatinine (UPC) ratio >= 1.0 at screening OR
  * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating. Refuse the use of effective means of contraception (men and women) in subjects of child-bearing potential

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Ghiaseddin A, Reardon D, Massey W, Mannerino A, Lipp ES, Herndon JE 2nd, McSherry F, Desjardins A, Randazzo D, Friedman HS, Peters KB. Phase II Study of Bevacizumab and Vorinostat for Patients with Recurrent World Health Organization Grade 4 Malignant Glioma. Oncologist. 2018 Feb;23(2):157-e21. doi: 10.1634/theoncologist.2017-0501. Epub 2017 Nov 13. PMID 29133513
- See also: Link to the Preston Robert Tisch Brain Tumor Center — http://www.cancer.duke.edu/btc/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/
- See also: Duke Cancer Center - Patient Care — http://www.dukehealth.org/cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants signed consent. 8 participants are considered screen failures. 40 participants received treatment.
Period: Overall Study
Arm/Group | Vorinostat & Bevacizumab
Started | 40
Completed | 38 (Participants who discontinued study drug for any reason.)
Not Completed | 2
Not completed — Still Receiving Treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Six-month Progression-free Survival (PFS6)
Description: The percentage of participants alive and progression-free at 6 months after the start of study treatment will be determined. Based on Response Assessment in Neuro-Oncology (RANO) criteria, progression is defined as a ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions; significant increase in T2/FLAIR; any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor; failure to return for evaluation as a result of death or deteriorating condition; or clear progression of non-measurable disease. PFS6 will be calculated from the date study treatment started until the date of progression or death, or the date of last follow-up if participants are alive without progression. Kaplan-Meier methods will be used to estimate survival.
Time Frame: 6 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 30 [16.8 to 44.4]

2. Secondary Outcome: Radiographic Response
Description: The percentage of participants with a complete or partial response as determined by modified Response Assessment in Neuro-Oncology (RANO) criteria will be determined. Complete Response (CR) is defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses) and accompanied by a stable or improving neurologic examination. Partial Response (PR) is defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids and accompanied by a stable or improving neurologic examination. Tumor assessments are done at baseline and the end of every second cycle (every 8 weeks) thereafter.
Time Frame: 3 Years
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vorinostat & Bevacizumab: Patients will be administered bevacizumab every 2 weeks and vorinostat will be taken on days 1-7 and 15-21 of each 28-day cycle at 400 mg per day.
  Vorinostat
  Bevacizumab
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 22.5 [12.1 to 37.7]

3. Secondary Outcome: Percentage of Participants Who Experience Grade 3 or Greater, Treatment Related, Non-hematologic Toxicities.
Description: The percentage of participants who experience grade 3 or greater, treatment-related, non-hematologic toxicities will be calculated.
Time Frame: 2.7 Years
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 40

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time in months from the start of protocol treatment until the date of progression or death if death occurred before progression. If the participant is alive and progression-free, PFS will be censored at the date of last follow-up. Kaplan-Meier methods will be used to estimate progression-free survival.
Time Frame: 3 Years
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
months | 3.7 [2.9 to 4.8]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time in months from the start of protocol treatment until the date of death, or the date of last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: 3 Years
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat & Bevacizumab
Number analyzed (Participants) | 40
months | 10.4 [7.6 to 12.8]

ADVERSE EVENTS:
Time Frame: From the start of study treatment for a patient until 30 days after treatment is discontinued.
Description: Patients will be evaluated for adverse events (AEs) (all grades), serious AEs, and adverse events requiring study drug interruption or discontinuation at each study visit for the duration of their participation in the study.
Groups:
- Vorinostat & Bevacizumab: Patients will be evaluated for adverse events (all grades), serious adverse events, and adverse events requiring study drug interruption or discontinuation at each study visit for the duration of their participation in the study.
Arm/Group | Vorinostat & Bevacizumab
Serious Adverse Events (participants affected / at risk) | 12/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat & Bevacizumab (N=40)
Sinus bradycardia (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Malaise (General disorders) | 1
Lung infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Edema cerebral (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 7
Confusion (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat & Bevacizumab (N=40)
Anemia (Blood and lymphatic system disorders) | 15
Sinus bradycardia (Cardiac disorders) | 5
Ear pain (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 11
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 28
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 6
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 28
Pain (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 32
Neutrophil count decreased (Investigations) | 22
Platelet count decreased (Investigations) | 33
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 27
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 27
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 5
Dysphasia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 17
Memory impairment (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 2
Pyramidal tract syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 13
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 12
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 9
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 14
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes